CLINICAL TRIAL: NCT06074185
Title: Treating Respiratory Emergencies in Children Study
Acronym: T-RECS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Utah (Other); University at Buffalo (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Matt Hansen, Professor, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00138724
Record Dates: First submitted 2023-08-10; First posted 2023-10-10 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-02

CONDITIONS: Asthma in Children
MeSH Terms: interventions — Ipratropium; Dexamethasone

STUDY DESIGN:
Intervention Model Description: This is a before-and-after study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continue current care (No Intervention): In this arm, participants will be treated using the existing EMS protocol, and evaluate patient outcomes.
- Treatment bundle and checklist (Experimental): In this arm, we will implement a new treatment protocol with the study bundle, and evaluate patient outcomes.
  Interventions: Drug: Ipratropium Bromide

INTERVENTIONS:
Drug: Ipratropium Bromide — The study intervention involves implementing a treatment bundle that includes inhaled ipratropium bromide and dexamethasone.
  Other Names: dexamethasone
  Arms: Treatment bundle and checklist

SUMMARY:
Over 200,000 children have a 911 Emergency Medical Services (EMS) activation for respiratory distress each year, most of whom have acute wheezing. Early treatment in the prehospital setting could more rapidly relieve respiratory distress symptoms, prevent hypoxia, reduce invasive interventions, and reduce the need to be hospitalized, thereby facilitating earlier return to normal daily activities. Preliminary data from one site found hospital admission was reduced from 30% to 21% among children when an EMS system introduced a pediatric asthma protocol with oral dexamethasone. The current standard for Emergency Department (ED) treatment for acute wheezing for children two and older includes inhaled ipratropium and dexamethasone. These treatments have a longstanding history of safety and are effective in preventing hospitalization when used early in the ED. Specific treatment protocols generally direct prehospital care. Ipratropium and dexamethasone are recommended by national EMS organizations that develop model protocols for prehospital care. However, only 25% of EMS agencies from large US metropolitan areas allow ipratropium, and only 10% include dexamethasone in their treatment protocols. A clinical trial is critically needed to evaluate whether the significant EMS resources required to implement interventions for children with life-threatening wheezing that have proven benefit in the ED result in improved patient outcomes. The overall objective of this three-site pilot trial is to address specific questions related to the implementation of the study and ensure its feasibility. The study will be conducted in the Pediatric Emergency Care Applied Research Network (PECARN) EMS Affiliates (EMSAs). The investigators will include patients aged 2-17 who have a 911 call for acute life-threatening wheezing. The specific aims are 1) to develop and produce a prehospital checklist for the treatment bundle, including ipratropium and dexamethasone, 2) to determine the feasibility of collecting patient outcomes for wheezing children treated in the EMS system, and 3) to evaluate the implementation of the EMS treatment bundle and checklist using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework. Our overall hypothesis is that the study will be feasible to implement. This study will provide the necessary data to ensure the eventual trial is feasible, primarily by establishing the ability to measure the outcomes of interest as well as evaluating implementation. This study is innovative by focusing on pediatric care in the prehospital environment, a critical component of our emergency care system that is often neglected in research.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 2-17 years; AND
2. Transported by EMS through 911 activation; AND
3. Prior history of wheeze/asthma, current asthma symptoms (dyspnea or wheeze); AND
4. At least 4 of the following:

   * Visible use of accessory muscles/retractions
   * Inspiratory and expiratory wheezing or silent chest
   * Abnormal respiratory rate for age

     * For < 6 years ≥ 46 breaths/min
     * For ≥ 6 years ≥ 36 breaths/min
   * Agitation, drowsiness, or confusion
   * Oxygen saturation < 93% on room air

Exclusion Criteria:

1. History of albuterol, ipratropium, or dexamethasone allergy
2. Known or suspected pregnancy
3. Prisoner
4. Croup
5. Suspected airway foreign body
6. Respiratory distress not due to bronchospasm/wheeze
7. Parent, legally authorized representative (LAR), subject, and/or family member objects to participation prior to treatment

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients admitted to the hospital in each group | Within 24 hours of the index EMS encounter
  Whether or not the patient was admitted to the hospital after the index EMS encounter

SECONDARY OUTCOMES:
NIH Patient-Reported Outcomes Measurement Information Systems (PROMIS) asthma impact scale | 6-8 days after the index EMS encounter
  Quality of life score for asthma. Range 0-100. A higher score equates to poorer quality of life.

OTHER OUTCOMES:
Rate of successful primary and secondary outcome measurement among participants | Through 8 days after enrollment
  We will evaluate the feasibility of collecting the main study outcomes among study participants
Proportion of patients who require a critical care intervention | Within one week of the index EMS encounter
  Use of bag mask ventilation, non-invasive positive pressure ventilation, endotracheal intubation, high-flow nasal cannula, Extra Corporeal Membrane Oxygenation (ECMO), and Cardio Pulmonary Resuscitation (CPR)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L Hansen, MD, MCR, Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (3):
  - University at Buffalo, Buffalo, New York
  - Mecklenburg County EMS, Charlotte, North Carolina
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No